CLINICAL TRIAL: NCT05224986
Title: Lifestyle Patterns and Glycemic Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Associate Professor of Nutritional Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAT8914; R01DK128154 (NIH)
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: A randomized, parallel-arm clinical intervention study to assess the role of variability in lifestyle behaviors on glucose control and body composition in adults with pre-diabetes. The goal is to test whether following a fixed schedule improves glucose control and insulin sensitivity and reduces adiposity compared to those who maintain a variable schedule.
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded to the intervention or purpose of the study but will be told that rest-activity patterns will be examined in the context of well-being and that we will test the influence of these lifestyle patterns on glucose control and body composition. Although the investigators and research assistant directly involved in the conduct of the study cannot be blinded to participant assignment to the intervention or control group, the technicians involved in sample processing and the biostatistician (Dr. Cheng) will be blinded to this information to reduce the risk of bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Variable Schedule (No Intervention): Participants randomized to Variable Schedule (VS) will be asked to maintain their usual habits for 12 weeks.
- Fixed Schedule (Experimental): Participants randomized to Fixed Schedule (FS) will be asked to stabilize their lifestyle behaviors for 12 weeks.
  Interventions: Behavioral: Fixed Schedule

INTERVENTIONS:
Behavioral: Fixed Schedule — Participants will be asked to maintain a fixed schedule for 12 weeks.
  Arms: Fixed Schedule

SUMMARY:
The goal of the proposed study is to evaluate the feasibility and initial efficacy of stabilizing lifestyle behaviors to improve glucose control and body composition in patients with pre-diabetes.

The investigator proposes that following stable lifestyle behaviors will improve patients' glucose control, body composition, and liver fat. The results from this study has the potential to impact clinical practice and patient care.

DETAILED DESCRIPTION:
Variability in lifestyle behaviors has been associated with adverse health, specifically poor glucose control. The project proposes to test whether reducing this variability improves glycemia in patients with pre-diabetes. If successful, this simple positive lifestyle message to keep stable behaviors has the potential to improve the health of millions of adults worldwide.

This project will enroll participants with pre-diabetes who have erratic lifestyle behaviors and randomize them to either maintain their usual habits (control group) or stabilize their behaviors (stability group). Both groups will be followed for 12 weeks. Before the start of the 12-week period, all participants will track their sleep for 2 weeks and will wear a glucose monitor to measure their glucose levels. At the start and end of the 12-week period, they will come to the research lab to undergo a glucose tolerance test. This test will measure how their body reacts to a glucose load. They will also undergo magnetic resonance imaging and spectroscopy scanning. This scan will provide information on body composition and liver fat content.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetic kg/m2 (hemoglobin A1c 5.7-6.9%)
* 25 years or older
* BMI between 25-39.9 kg/m2
* Sleep duration ≥6 hours a night assessed with wrist actigraphy (for 14 nights)
* Variable bedtime, SD≥45 minutes.

Exclusion Criteria:

* Chronic Kidney Disease (GFR<60)
* Uncontrolled hypertension (≥160/100 mmHg)
* Obstructive Sleep Apnea
* Psychiatric or neurological disorder
* Prevalent cardiovascular disease
* Dyslipidemia (triglycerides≥200 mg/dL)
* Medications that affect insulin sensitivity, glucose concentrations, and body weight
* Non-day or rotating shift workers
* Travel across time zones
* Active participation in weight loss program or within past 3 months
* Current or past alcohol/drug abuse

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Adipose Tissue Measurement - Total | 12 weeks
  Measuring total adiposity. Measured by MRI, includes both subcutaneous and visceral adipose tissue.
Adipose Tissue Measurement - Subcutaneous | 12 weeks
  Measurement of subcutaneous adiposity using MRI.
Adipose Tissue Measurement - Visceral | 12 weeks
  Measurement of visceral adiposity using MRI.
Glucose Area Under Curve | 12 weeks
  Testing glycemic control.The primary outcome variable is glucose under the curve during the oral glucose tolerance test.
Mean Amplitude of Glycemic Excursion and Standard Deviation of Mean Glucose | 12 weeks
  Testing glucose variability. The primary outcome variables are mean amplitude of glucose excursion and standard deviation of average glucose.

SECONDARY OUTCOMES:
Liver Fat Content | 12 weeks
  This is to assess liver fat measured by MRS and MRI in %.
Disposition Index | 12 weeks
  This is to assess disposition index, measured using HOMA-IR. The disposition index is the product of the insulogenic index and homeostatic model of assessment for insulin resistance.
Short-term Change in Glycemia | Baseline, up to 12 weeks
  Assessing whether short-term glycemia is changed by measuring fructosamine using two-sample t-tests.
Endothelial cell inflammation (sub-set, n≤10) | Baseline, 12 weeks
  NF-κB nuclear fluorescence area for pilot study.
White blood cells | Baseline, 12 weeks
  Leukocytes and neutrophils
Long-term Change in Glycemia | Baseline, 12 weeks
  Assessing whether long-term glycemia is changed by measuring hemoglobin A1c using two-sample t-tests.
Endothelial cell oxidative stress (sub-set, n≤10) | Baseline, 12 weeks
  redox sensitive fluorogenic probe fluorescence intensity for pilot study.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, Principal Investigator — Columbia University; Blandine Laferrere, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No